CLINICAL TRIAL: NCT04238533
Title: Enhanced Auto-Diagnostic Adaptive Precision Trainer for Myoelectric Prosthetic Users
Acronym: eADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: Design Interactive, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00041255; CDMRP-CDMRP OP160046 (Other: Department of Defense (per award terms))
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Amputation
Keywords: transradial; upper extremity; amputee; forearm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eADAPT (Active Comparator): This arm includes transradial amputees who will be assessed while using the eADAPT trainer.
  Interventions: Other: eADAPT training
- Conventional program (Active Comparator): This arm includes transradial amputees who will be assessed while using the conventional training program.
  Interventions: Other: Conventional training

INTERVENTIONS:
Other: eADAPT training — eADAPT training for myoelectric prosthesis users is the comparator training.
  Arms: eADAPT
Other: Conventional training — Conventional training with Myoboy has been the only training available to users.
  Arms: Conventional program

SUMMARY:
The eADAPT training consists of a variety of mobile games played on a mobile app (phone or tablet). A band is worn on the residual limb. Participants use muscle activation to send signals to execute certain movements in the game.

DETAILED DESCRIPTION:
Myoelectric prostheses provide upper limb movement control using electromyography (EMG) electrodes on the residual muscles to control arm and hand movements. Within the current generation of advanced prostheses, research has shown that most amputees rely on assistive devices rather than prostheses (27 - 54% use prostheses), and many users do not use all available features or stop using the device altogether. Part of the difficulty in learning to control upper limb myoelectric prostheses stems from the sequences of muscle inputs required to choose grips and modes, and move the limb.

Myoelectric prosthetic limbs can aide in regaining lost capabilities, but require intensive training to effectively operate. Learning to use a myoelectric prosthesis involves significant motor cortex plasticity and learning how to consciously control muscle contraction, level of activation, and isolation through repetitive exercises. The need to concentrate and continuously react during training is expected to decrease with use, but often takes amputees many months, with the result being that many users abandon the prosthesis before mastery is achieved.

Difficult training has been identified as a primary reason for low user acceptance.

Current training methods and tools can be expensive, are limited in their activation sites, transferability, and personalized training capabilities. Current one-size-fits-all training cannot be personalized for the patient, thereby ignoring or being unresponsive to their learning ability. This limitation factor reduces the level of acute positive patient outcomes that can be achieved. A need therefore exists for myoelectric training tools that are affordable, reliable, support conventional and state-of-the-art control schemes, adaptable to various patient needs, can improve patient clinical outcomes, motivate patients to train, and be used in the clinic and remotely by the patient.

To fill the identified gaps in myoelectric training tools, Design Interactive, Inc. (DI) developed a prototype of the Auto Diagnostic Adaptive Precision Trainer for Myoelectric Prosthesis users (ADAPT-MP), an adaptive, game-based modular software solution paired with an innovative, mobile hardware solution to support the upper limb prosthesis training continuum, including basic pre-prosthetic training through advanced skill training using the prosthesis.

Rationale Current prosthetic training is monotonous, expensive, specific to certain devices, and often cannot be brought home. The eADAPT-MP system has multiple engaging games of varying levels of difficulty, is inexpensive, is designed to be manufacturer and device agnostic, and is a tool users can bring with them almost anywhere. The upper limb amputee patient population would benefit from having a powerful telerehabilitation tool that is engaging and encourages prosthetic training to reduce abandonment of myoelectric prostheses and promote usability of myoelectric arms. However, there is a lack of randomized, controlled clinical data supporting myoprosthetic training on functional outcomes. Previously published clinical research on the effect of pre-prosthetic training on amputee health outcomes is represented by small, uncontrolled case studies, or the reliance on non-amputee participants.

ELIGIBILITY:
Inclusion Criteria:

* Amputation or missing limb at or above the wrist and below the elbow (transradial)
* Current myoelectric prosthesis user
* Sufficient neurological and cognitive function to operate the prosthesis effectively as assessed by research personnel during initial interviews;
* Sufficient neurological and cognitive function to operate a mobile device (phone, tablet) effectively;
* The patient is free of comorbidities that could interfere with the function of the prosthesis;
* Functional evaluation indicates that with training, use of a myoelectric prosthesis is likely to meet the functional needs of the individual when performing activities of daily living
* Age 18-70 years
* Able to independently read, speak and understand English for the purpose of consent, following instructions and completing surveys

Exclusion Criteria:

* Amputation or missing limb at a level that is not above the wrist and below the elbow (transradial)

  * Not currently a myoelectric user
  * Insufficient neurological and cognitive function to operate the prosthesis effectively as assessed by research personnel during initial interviews;
  * Insufficient neurological and cognitive function to operate a mobile device (phone, tablet) effectively
  * The patient has comorbidities that could interfere with function of the prosthesis;
  * Functional evaluation indicates that despite training, use of a myoelectric prosthesis is unlikely to meet the functional needs of the individual when performing activities of daily living;
  * Age <18 or >70 years
  * Participants with significant cognitive deficits or visual impairment that would preclude them from giving informed consent or following instructions during the study procedure, or the ability to obtain relevant user feedback.
  * Unable to independently read, speak and understand English for the purpose of consent, following instructions, and completing surveys

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Compliance | 3 weeks
  Compliance with the respective training protocol. For conventional exercise, patients will be contacted by phone once per week and asked if they were compliant with the training protocol. For the experimental (eADAPT) training protocol, utilization time will be recorded via the app and available for download for analysis. The difference in compliance between the two protocols will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Highsmith, PhD, Principal Investigator — University of South Florida
Locations (1):
- James A Haley VA, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No